CLINICAL TRIAL: NCT00420394
Title: Phase II Study of Preoperative Chemotherapy and Postoperative Chemo-Radiation for Newly Diagnosed, Potentially Resectable Gastric Cancer
Brief Title: Perioperative Chemoradiotherapy for Potentially Resectable Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOR446006ctil
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2007-06-20 (Estimated); Status verified 2007-01

CONDITIONS: Stomach Neoplasms
Keywords: Neoadjuvant chemotherapy; Adjuvant chemoradiotherapy; Adenocarcinoma of stomach and gastroesophageal junction
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Chemotherapy
Procedure: surgery
Procedure: radiotherapy

SUMMARY:
Rationale: Adjuvant chemoradiation considered as standard of care after curative surgery for adenocarcinoma of stomach and gastroesophageal cancer. Preoperative chemotherapy in the in locally advanced gastric cancer results in significant tumoral downstaging with improved rate of curative resections.

Purpose: To evaluate feasibility and safety of combination of preoperative chemotherapy and postoperative chemoradiation for locally advanced adenocarcinoma of stomach and gastroesophageal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed primary adenocarcinoma, poorly differentiated carcinoma, or carcinoma not otherwise specified, of stomach or gastro-esophageal junction.
2. T2-4 N0-3 M0. T1 tumors are eligible if T1N1-3
3. Disease must be clinically limited to the stomach or GEJ.
4. Pre-treatment Port-a-Cath insertion obligatory
5. No prior chemotherapy.
6. No prior radiotherapy.
7. Patients must be surgical candidates as determined by the treating surgeon.
8. Adequate organ function defined as:
9. Patients must have an ECOG Performance Status < 1.
10. Patients must be able to sign the informed consent document.

Exclusion Criteria:

1. Tis (in-situ carcinoma) and tumors determined to be TIN0 following endoscopy, endoscopic ultrasound and CT scanning.
2. Patients with primary carcinomas of the esophagus.
3. Prior chest or upper abdomen radiotherapy, prior systemic chemotherapy within the past 5 years, or prior esophageal or gastric surgery.
4. Patients with evidence of metastatic disease are not eligible.
5. New York Heart Association Class III or IV heart disease.
6. Severe co-morbid conditions or nonmalignant illness whose control may be jeopardized by complications of the study treatment.
7. Pregnant or lactating women or men unable or unwilling to practice contraception are excluded.
8. Any history of prior malignancy (other than non-melanoma skin cancer, in-situ cervical cancer, or superficial transitional cell bladder cancer).
9. Clinically significant hearing loss.
10. Patients with a history of seizure disorder who are receiving phenytoin, phenobarbital, or other antiepileptic medication.
11. Patients who cannot fully comprehend the therapeutic implications of the protocol or comply with its requirements.
12. Patients with any medical or psychiatric condition or disease which, in the investigator's judgment, would make the patient inappropriate for entry into this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-04

PRIMARY OUTCOMES:
Feasibility of the study regimen.

SECONDARY OUTCOMES:
Rate of R0 resection following chemotherapy.
Morbidity and mortality of surgery following chemotherapy.
Overall and progression free survival following the study treatment plan

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Tokar, MD, Study Chair — Soroka University Medical Center and Ben-Gurion University of the Negev
Locations (1):
- Soroka University Medical Center,Oncology Center, Beersheba, Israel